CLINICAL TRIAL: NCT01035203
Title: Effects of a Brief Endurance Exercise Program and of a Cognitive Behavioural Therapy on Patients With Cancer-related Fatigue
Brief Title: Exercise Versus Cognitive Behavioural Therapy on Cancer-related Fatigue
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Fernando Dimeo, MD, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 176-25/kmo
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Fatigue; Mood; Maximal Oxygen Uptake
MeSH Terms: conditions — Fatigue | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioural therapy (Active Comparator)
  Interventions: Behavioral: Cognitive behavioural therapy
- Exercise (Experimental): Endurance training (walking on a treadmill) 3 x weekly for 4 weeks
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Endurance exercise 3 times weekly for 45 minutes, 4 weeks long
  Arms: Exercise
Behavioral: Cognitive behavioural therapy — Teaching of techniques to reduce fatigue and to improve stamina
  Arms: Cognitive behavioural therapy

SUMMARY:
The investigators compare the effects of two interventions, an endurance exercise program and a cognitive behavioural therapy, on the fatigue, quality of life, mood and physical performance of patients with a cancer-related fatigue syndrome. The intervention will be carried out for 4 weeks. Tests will be carried out at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Histologically confirmed neoplastic disease
* Treatment (chemotherapy or radiation) completed.
* No treatment in the previous 4 weeks
* Ability to understand written German

Exclusion Criteria:

* Health conditions which can be aggravated by exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-07 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Fatigue scores on the Brief Fatigue Inventory (BFI) | 4 weeks

SECONDARY OUTCOMES:
Maximal oxygen uptake (VO2max) on a treadmill stress test. | 4 weeks
Scores on the HADS (Hospital Anxiety and Depression Scale) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Berlin, State of Berlin, Germany